CLINICAL TRIAL: NCT00571961
Title: Pharmacokinetic Interactions Between Buprenorphine and Kaletra (Lopinavir/Ritonavir)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, R. Douglas Bruce, MD, MA, Assistant Professor of Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0511000791; M118687
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: HIV; Pharmacokinetics; Buprenorphine; Kaletra; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir; Buprenorphine; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HIV negative subjects currently enrolled in a long-term buprenorphine maintenance therapy program for at least 3 months who have been on stable dose of buprenorphine for at least 3 weeks will be admitted to the General Clinical Research Center (GCRC) for pharmacokinetic (PK) blood draws at intervals over a 24-hour period. Subjects will then receive Kaletra and buprenorphine coadministered for 14 days. Subjects will be admitted to the GCRC for a second PK sampling day.
  Interventions: Drug: Kaletra (lopinavir/ritonavir); Drug: buprenorphine; Other: Clinical evaluations/Blood draws

INTERVENTIONS:
Drug: Kaletra (lopinavir/ritonavir) — 4 tablets, once a day (800 mg/dose) on Days 2 through 14 of this study
Drug: buprenorphine — Buprenorphine will be obtained through prescription at the subject's drug treatment program.
Other: Clinical evaluations/Blood draws — Physical examinations, vital sign measurements, 12-lead electrocardiogram (ECG), clinical laboratory evaluations (blood chemistry and blood counts), PK blood draws.

SUMMARY:
The main purpose of this protocol is to study the effect of an HIV medication, Kaletra (lopinavir/ritonavir), on buprenorphine in non-HIV infected people who have been receiving the same dose of buprenorphine for at least 3 weeks.

Study Hypothesis:

Kaletra (lopinavir/ritonavir) will increase buprenorphine plasma levels without any significant clinical effect on the subject or need for dose adjustment.

DETAILED DESCRIPTION:
Buprenorphine (BUP) is a partial opiate agonist dosed sublingually for both supervised opiate withdrawal and maintenance for opiate dependence. Until recently, methadone has been the mainstay of pharmacological treatment for opiate-dependent persons with HIV infection. In October, 2002, buprenorphine (BUP) was approved for opiate maintenance and can be prescribed by primary care physicians. It is anticipated that many HIV specialists will begin prescribing BUP for their HIV+ patients on ARVs with a history of opiate dependence. This will continue to increase in importance as a method of treatment for this patient population for the following reasons: 1) Multiple federal programs are working to encourage the use of BUP in primary care, especially HIV primary care, settings. The goal of these programs is to increase opiate treatment slots across the country. 2) Many methadone programs have wait lists or regulations (e.g., daily dosing) which may not be possible for some patients. BUP, with its flexibility in dosing and ease of use, will increasingly become a first line in the treatment of opioid dependence.

Buprenorphine administration carries the theoretical risk of drug interactions with respect to both inhibition or induction of BUP as well as similar effects on medications co-administered with BUP. Interactions may lead to under or overdosing of buprenorphine and/or antiretroviral agents with resultant adverse clinical consequences.

Buprenorphine's effects on Kaletra and other ARVs cannot be predicted based on prior experience with methadone because BUP metabolism appears to differ from methadone in terms of its substrate and effects on cytochrome P450.

Limited information currently exists regarding interactions between HIV therapeutic agents and buprenorphine. Similar to buprenorphine, the protease inhibitors, and NNRTIs are metabolized primarily via the CYP3A4 isozyme of the cytochrome P450 system. The extent to which methadone levels decrease with induction of cytochrome P450 isoenzymes has been correlated clinically with severity of symptoms of withdrawal. Similar studies with buprenorphine are not yet available. Interactions between buprenorphine and antiretroviral agents may complicate the management of HIV disease when these medications are coadministered. In a small sample study, there was no increase in buprenorphine dosing required when co-administered with Sustiva. However, in one study with liver microsomes, ritonavir inhibited the metabolism of buprenorphine at CYP 3A4, but the clinical significance of this inhibition could not be demonstrated. It is well known that in vitro and in vivo studies do not fully correlate with one another and empiric pharmacologic interaction studies in human subjects are necessary.

The treatment of opiate addiction is a complicated and labor intensive practice. This study will require the use of Kaletra alone in HIV negative opiate dependent patients. This is critical to ascertain the reality of both objective data (levels of buprenorphine and lopinavir), as well as valid subjective symptoms of opiate withdrawal (symptoms that addicts have previously experienced and can more readily communicate).

ELIGIBILITY:
Inclusion Criteria:

* Chronic BUP users enrolled in BUP program, receiving BUP for at least 3 months and on a stable BUP dose for at least 3 weeks.
* Acceptable medical history, physical examination, 12 lead electrocardiogram, and clinical laboratory evaluations consistent with BUP maintenance
* Subjects who meet the criteria of opiate dependence, are enrolled in long-term BUP maintenance therapy, and have been on a stable dose of BUP for at least 3 weeks.
* Body weight >60 kg for males and >40 kg for females
* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2.
* Male or females, ages 18 to 65 years.
* Women of childbearing potential (WOCBP) must not be nursing, pregnant and on adequate non-hormonal contraception to avoid pregnancy. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Study Day 1.

Exclusion Criteria:

Sex and Reproductive Status Exceptions

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks before and after the study.
* WOCBP using a prohibited contraceptive method (oral, injectable, or implantable hormonal agents)
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration.

Medical History and Concurrent Diseases

* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* History of nephrolithiasis
* History of acute or chronic pancreatitis.
* History of uncontrolled chronic medical illness which could adversely affect the subject's adherence to study protocol or affect patient safety in the opinion of the investigator
* Use of any medication thought to significantly alter the metabolism of Kaletra, Buprenorphine or naloxone.
* History of any hemolytic disorders (including drug-induced hemolysis).
* Proven or suspected acute hepatitis at the time of study entry.
* Current or recent (within 3 months) gastrointestinal disease which would interfere with the conduct or interpretation of the study.
* Any major surgery within 4 weeks of enrollment. Minor surgical procedures requiring local anesthesia are exceptions.
* Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of enrollment.
* Blood transfusion within 4 weeks of enrollment.
* Inability to tolerate oral medication.
* Inability to tolerate venipuncture and/or absence of secure venous access.
* Inability to refrain from smoking during in-patient period
* Known or suspected HIV infection (subjects who are found to be positive upon screen for HIV will be excluded).
* Known active drug or alcohol abuse, which in the opinion of the investigator makes study participation to completion unlikely.
* Any other sound medical, psychiatric and/or social reason as determined by the Investigator.

Physical and Laboratory Test Findings

* Evidence of organ dysfunction or any clinically relevant deviations from the norms observed in a buprenorphine treated population in physical examination, vital signs, ECG or clinical laboratory determinations.
* Ingestion of alcohol within 24 hours prior to the dose of study medication
* Positive breathalyzer alcohol test, or positive urine screen for barbiturates, benzodiazepines, amphetamines or opiates other than buprenorphine.
* Positive blood screen for HIV antibody.
* QTc interval >450 msec for males or >470 msec for females.
* Second or third-degree AV block.
* Creatinine clearance(as estimated by method of Cockcroft and Gault) less than 80 mL/min.
* CLcr=0.85(females only)x(140-age)x weight(kg)
* serum creatinine(mg/dL)x 72
* Subjects with bilirubin >2 mg/dL, serum albumin <2.5 g/dL and ascites, AST and ALT >3 times ULN, hemoglobin <9 g/dL, and platelet count <75,000/mm3.
* Positive serum or urine for HCG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Bruce, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Result] Bruce RD, Altice FL, Moody DE, Morse GD, Andrews L, Lin SN, Fang WB, Ma Q, Friedland GH. Pharmacokinetic interactions between buprenorphine/naloxone and once-daily lopinavir/ritonavir. J Acquir Immune Defic Syndr. 2010 Aug;54(5):511-4. doi: 10.1097/qai.0b013e3181d3cad3. PMID 20672450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV negative subjects currently enrolled in a long-term buprenorphine maintenance therapy program for at least 3 months who have been on stable dose of buprenorphine/naloxone (BUP/NLX) for at least 3 weeks will be admitted to the General Clinical Research Center (GCRC) for pharmacokinetic (PK) blood draws at intervals over a 24-hour period.
Pre-assignment Details: Once admitted to the GCRC, subjects were maintained on 16 mg of BUP/NLX daily, except for 1 patient on 24 mg. As baseline, subjects on steady-state BUP/NLX were hospitalized and underwent pharmacokinetic investigation over a 24-hr period. Subjects served as their own controls.
Groups:
- Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg: Subjects received 800mg/200mg of LPV/r once daily in addition to BUP/NLX that the subjects were already being previously maintained on. These drugs were coadministered for a minimum of 10 days under direct observation.
Period: Overall Study
Arm/Group | Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg: Subjects received 800mg/200mg of LPV/r in addition to BUP/NLX that the subjects were already being previously maintained on. These drugs were coadministered for a minimum of 10 days under direct observation.
Arm/Group | Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg
Number analyzed (Participants) | 12
Age Continuous [Median (Full Range); unit: years] | 42 (1) [29 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Area Under the Curve With LPV/r (ng/mL*hr)
Description: Pharmacokinetic parameters were determined by use of non compartmental methods. The area under the plasma concentration versus time curve was determined by use of the trapezoidal rule and measured over a 24-hr time period.
Time Frame: 15 days
Measure: Mean (Standard Deviation); unit: (ng/mL)*hr
Arm/Group | Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg
Number analyzed (Participants) | 12
(ng/mL)*hr | 46.2 (15.3)

ADVERSE EVENTS:
Arm/Group | Lopinavir Coformulated With Ritonavir (LPV/r), 800mg/200mg
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No